CLINICAL TRIAL: NCT01831544
Title: Multi Center, Prospective, Non-Randomized, Single-Arm Trial Evaluating the Clinical Safety and Performance Of the HeartWare MVAD® System For the Treatment of Advanced Heart Failure
Brief Title: A Clinical Trial to Evaluate the HeartWare MVAD® System (MVAdvantage)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment terminated due to higher rate of thrombosis events than expected.
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HW-MVAD-01
Record Dates: First submitted 2013-04-08; First posted 2013-04-15 (Estimated); Results first posted 2020-04-07 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2022-07

CONDITIONS: Heart Failure
Keywords: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MVAD® Pump (Experimental): Implant of HeartWare MVAD® System
  Interventions: Device: HeartWare MVAD® System

INTERVENTIONS:
Device: HeartWare MVAD® System — The HeartWare MVAD® System consists of a small, wearless, continuous flow pump and associated surgical tools and implant accessories, peripheral components which control and power the system, and a monitor which allows for programming and monitoring of the system

SUMMARY:
This multi-center, prospective, non-randomized, single-arm trial will investigate the safety and performance of the HeartWare® Miniaturized Ventricular Assist Device (MVAD®) system over 24 months in subjects with advanced heart failure

DETAILED DESCRIPTION:
This multi-center, prospective, non-randomized, single-arm trial will investigate the safety and performance of the Miniaturized Ventricular Assist Device (MVAD®) system over 24 months in subjects with advanced heart failure. The primary endpoint is survival at 6 months presented as a simple proportion (subjects alive on the MVAD® pump divided by endpoint eligible subjects). Secondary endpoints include the incidence of bleeding, incidence of major infections (per INTERMACS definitions), time to death, incidence of all device failures and device malfunctions, Health Status improvement, and Functional status improvement. Safety measures will include the frequency and rates of adverse events, overall and for each specific event, which will be collected throughout VAD support.

ELIGIBILITY:
Inclusion Criteria:

1. Must be ≥18 years of age at consent
2. Subjects with advanced heart failure symptoms (Class IIIB or IV) who meet one of the following):

   1. on optimal medical management including dietary salt restriction and diuretics, for at least 45 out of the last 60 days and are failing to respond; or
   2. in Class III or Class IV heart failure for at least 14 days and dependent on intra-aortic balloon pump (IABP) and/or inotropes.
3. Left ventricular ejection fraction ≤25%.
4. Female subjects of childbearing potential must agree to use adequate contraceptive precautions (defined as oral contraceptives, intrauterine devices, surgical contraceptives or a combination of condom and spermicide) for the duration of the study.
5. The subject has signed the informed consent form.

Exclusion Criteria:

1. Body Mass Index (BMI) > 47.
2. Body Surface Area (BSA) < 1.0 m2.
3. Partial or full mechanical circulatory support within thirty days of implant.
4. Existence of any ongoing mechanical circulatory support (MCS) other than an intra-aortic balloon pump (IABP) or TandemHeart PTVA®.
5. Prior cardiac transplant or cardiomyoplasty.
6. History of confirmed, untreated abdominal or thoracic aortic aneurysm (diameter > 5 cm).
7. Acute myocardial infarction within 14 days of implant as diagnosed by ST or T wave changes on the electrocardiogram (ECG), diagnostic biomarkers, ongoing pain and hemodynamic abnormalities.
8. On ventilator support for > 72 hours within the four days immediately prior to implant.
9. Pulmonary embolus within three weeks of implant as documented by computed tomography (CT) scan or nuclear scan.
10. Symptomatic cerebrovascular disease, stroke within 180 days of implant or > 80% stenosis of carotid or cranial vessels in the absence of confirmed collateral circulation
11. Uncorrected moderate to severe aortic insufficiency.
12. Severe right ventricular failure as defined by the anticipated need for extracorporeal membrane oxygenation (ECMO) at the time of screening.
13. Active, uncontrolled infection diagnosed by a combination of clinical symptoms and laboratory testing, including but not limited to, continued positive cultures, elevated temperature and white blood cell (WBC) count, hypotension, tachycardia, generalized malaise despite appropriate antibiotic, antiviral or antifungal treatment.
14. Uncorrected thrombocytopenia or generalized coagulopathy (e.g., platelet count < 75,000, International Normalized Ratio (INR) > 2.0 or Partial Thromboplastin Time (PTT) > 2.5 times control in the absence of anticoagulation therapy).
15. Intolerance to anticoagulant or antiplatelet therapies or any other peri- or postoperative therapy that the investigator may administer based upon the subject's health status.
16. Serum creatinine > 3.0 mg/dL within 72 hours of implant or requiring dialysis.
17. Specific liver enzymes [Aspartate Aminotransferase (AST) (SGOT), and Alanine Aminotransferase (ALT) (SGPT)] > 3 times upper limit of normal within 72 hours of implant.
18. A total bilirubin > 3 mg/dL within 72 hours of implant, or biopsy proven liver cirrhosis or portal hypertension.
19. Pulmonary vascular resistance (PVR) is demonstrated to be unresponsive to pharmacological manipulation.
20. Subjects with a mechanical heart valve.
21. Etiology of heart failure is due to, or associated with, uncorrected thyroid disease, obstructive cardiomyopathy, pericardial disease, amyloidosis, active myocarditis or restrictive cardiomyopathy.
22. History of severe COPD or severe restrictive lung disease (e.g. FEV1 < 50% predicted value).
23. Participation in any other trial involving investigational drugs or devices within 4 weeks prior to screening and last visit of the trial.
24. Severe illness, other than heart disease, which would limit survival to < 3 years.
25. Peripheral vascular disease with rest pain or ischemic ulcers of the extremities.
26. Pregnancy and breast feeding.
27. Psychiatric disease, irreversible cognitive dysfunction or psychosocial issues that are likely to impair compliance with the CIP and LVAD.
28. Subject unwilling or unable to comply with trial requirements.
29. Technical obstacles, which pose an inordinately high surgical risk, in the judgment of the investigator.
30. Employees of the investigator or trial site, with direct involvement in this trial or other trials under the direction of the investigator or trial site, as well as family members or employees of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2015-07-14 (Actual); Primary Completion 2015-09-01 (Actual); Study Completion 2017-02-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Schueler, Principal Investigator — Freeman Hospital Newcastle Hospitals NHS Foundation Trust
Locations (11):
- St. Vincents Hospital, Darlinghurst, Australia
- Medical University AKH Vienna, Vienna, Austria
- Hospitalier Pitié-Salpétrière, Paris, France
- Germany (6):
  - The Heart and Diabetes Center NRW, Bad Oeynhausen
  - German Heart Institute Berlin DHZB, Berlin
  - Duesseldorf University Hospital, Düsseldorf
  - Uniklinik Hamburg Eppendorf (UKE), Hamburg
  - Hannover Medical School MHH, Hanover
  - University of Leipzig Heart Center, Leipzig
- United Kingdom (2):
  - Freeman Hospital, Newcastle upon Tyne
  - Papworth Hospital NHS Foundation, Papworth Everard

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MVAD® Pump
Started | 11
Completed | 8
Not Completed | 3
Not completed — Death | 1
Not completed — Still on original MVAD device | 2

BASELINE CHARACTERISTICS:
Arm/Group | MVAD® Pump
Number analyzed (Participants) | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (14.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 11
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Austria | 2
  United Kingdom | 2
  Australia | 2
  Germany | 5
Height [Mean (Standard Deviation); unit: centimeters] | 177.3 (6.41)
Weight [Mean (Standard Deviation); unit: kilograms] | 73.5 (14.36)
Blood Pressure [Mean (Standard Deviation); unit: mmHg]
  Systolic | 101 (15.58)
  Diastolic | 65.9 (10.10)
Intermacs Patient Profile [Number; unit: participants]
  1 - Critical cardiogenic shock | 0
  2 - Progressive decline | 0
  3 - Inotrope dependent | 6
  4 - Resting symptoms | 5
  5 - Exertion intolerant | 0
  6 - Exertion limited | 0
  7 - Advanced NYHA III | 0
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 23.2 (3.41)
Body Surface Area [Mean (Standard Deviation); unit: m^2] | 1.9 (0.21)

OUTCOME MEASURES:

1. Primary Outcome: Survival
Description: Primary Endpoint: survival at 6 months presented as a simple proportion. Transplants, explants for recovery and exchanges (to a device other than the MVAD® pump) prior to 6 month follow-up will be eligible for endpoint analysis, with survival status identified at the time of procedure.
Time Frame: Six month
Measure: Count of Participants; unit: Participants
Arm/Group | MVAD® Pump
Number analyzed (Participants) | 11
Participants | 10

2. Secondary Outcome: Survival
Description: Survival at 24 months presented as a simple proportion. Transplants, explants for recovery and exchanges (to a device other than the MVAD® pump) prior to 24 month follow-up will be eligible for endpoint analysis, with survival status identified at the time of procedure.
Time Frame: Two years
Measure: Count of Participants; unit: Participants
Arm/Group | MVAD® Pump
Number analyzed (Participants) | 11
Participants | 10

3. Secondary Outcome: Survival: Number of Participants Who Died by Six Months and Two Years
Description: Survival: Number of participants who died by six months and two years
Time Frame: Six months and two years
Population: The number of subjects enrolled in the study and implanted with MVAD System
Measure: Count of Participants; unit: Participants
Arm/Group | MVAD® Pump
Number analyzed (Participants) | 11
Participants
  Subjects who died by 6 months, cumulative | 1
  Subjects who died by 2 years, cumulative | 1

4. Secondary Outcome: Incidence of Major Bleeding
Description: Incidence of major bleeding, per INTERMACS definition
Time Frame: Six months and two years
Population: The number of subjects enrolled in the study and implanted with MVAD System.
Measure: Count of Participants; unit: Participants
Arm/Group | MVAD® Pump
Number analyzed (Participants) | 11
Participants
  Subjects who had an incidence of major bleeding by 6 months, cumulative | 5
  Subjects who had an incidence of major bleeding by 2 years, cumulative | 7

5. Secondary Outcome: Incidence of All Device Failures and Device Malfunctions
Description: Incidence of all device failures and device malfunctions per INTERMACS definition
Time Frame: Six months and two years
Population: The number of subjects enrolled in the study and implanted with MVAD System
Measure: Count of Participants; unit: Participants
Arm/Group | MVAD® Pump
Number analyzed (Participants) | 11
Participants
  Subjects with Device Malfunction by 6 months, cumulative | 5
  Subjects with Device Malfunction by 2 years, cumulative | 6

6. Secondary Outcome: Incidence of Major Infection
Description: Incidence of major infection, per INTERMACS definition
Time Frame: Six months and two years
Population: The number of subjects enrolled in the study and implanted with MVAD System.
Measure: Count of Participants; unit: Participants
Arm/Group | MVAD® Pump
Number analyzed (Participants) | 11
Participants
  Subjects with Major Infection by 6 months, cumulative | 3
  Subjects with Major Infection by 2 years, cumulative | 5

7. Secondary Outcome: Incidence of Neurological Dysfunction
Description: Incidence of neurological dysfunction per INTERMACS definition
Time Frame: Six months and two years
Population: The number of subjects enrolled in the study and implanted with MVAD System.
Measure: Count of Participants; unit: Participants
Arm/Group | MVAD® Pump
Number analyzed (Participants) | 11
Participants
  Subjects with Neurological Dysfunction by 6 months, cumulative | 0
  Subjects with Neurological Dysfunction by 2 years, cumulative | 0

8. Secondary Outcome: Health Status Change, as Measured by KCCQ and EuroQol EQ-5D-5L
Description: Health Status change, as measured by KCCQ and EuroQol EQ-5D-5L. Measured at baseline, 6 month visit and 24 month visit. Change from baseline at 6 month visit and 24 month visit were measured. The EQ-5D-5L overall score is between 0 and 1. 1 being the best score and 0 being the worst score. The KCCQ score is between 0 and 100. 100 being the best score and 0 being the worst score.
Time Frame: Six month and 24 month visit
Population: No data displayed because Outcome Measure has zero total participants analyzed
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | MVAD® Pump
Number analyzed (Participants) | 11
Score
  EQ5D Baseline | 0.63 (0.29)
  EQ5D 6 Months: number analyzed (Participants) | 7
  EQ5D 6 Months | 0.67 (0.34)
  EQ5D 6 Months vs baseline: number analyzed (Participants) | 7
  EQ5D 6 Months vs baseline | 0.13 (0.47)
  EQ5D at 24 Months: number analyzed (Participants) | 3
  EQ5D at 24 Months | 0.94 (0.11)
  EQ5D 24 Months vs baseline: number analyzed (Participants) | 3
  EQ5D 24 Months vs baseline | 0.21 (0.31)
  KCCQ Overall Score Baseline | 47.86 (21.79)
  KCCQ Overall Score 6 Months: number analyzed (Participants) | 7
  KCCQ Overall Score 6 Months | 72.63 (16.10)
  KCCQ Overall Score 6 Months vs Baseline: number analyzed (Participants) | 7
  KCCQ Overall Score 6 Months vs Baseline | 22.49 (31.16)
  KCCQ Overall Score 24 Months: number analyzed (Participants) | 3
  KCCQ Overall Score 24 Months | 81.94 (11.37)
  KCCQ Overall Score 24 Months vs Baseline: number analyzed (Participants) | 3
  KCCQ Overall Score 24 Months vs Baseline | 23.5 (35.15)

9. Secondary Outcome: Functional Status Change, as Measured 6-minute Walk
Description: Functional status change, as measured by 6-minute walk. Distance walked in meters in 6 minutes measured at baseline, 6 months and 24 month visit. Change from baseline at 6 month visit and 24 month visit were measured
Time Frame: 6 month and 24 month visit
Population: Subjects with implant attempt
Measure: Mean (Standard Deviation); unit: Distance in meters
Arm/Group | MVAD® Pump
Number analyzed (Participants) | 11
Distance in meters
  Baseline: number analyzed (Participants) | 10
  Baseline | 257.83 (93.7)
  6 month visit: number analyzed (Participants) | 5
  6 month visit | 445.4 (71.71)
  Change between 6 month visit and baseline: number analyzed (Participants) | 4
  Change between 6 month visit and baseline | 213 (81.97)
  2 year visit: number analyzed (Participants) | 2
  2 year visit | 402 (74.95)
  Change between 2 year visit and baseline: number analyzed (Participants) | 1
  Change between 2 year visit and baseline | 313 (0)

10. Secondary Outcome: Frequency and Rates of Adverse Events(AEs)
Description: Frequency and rates of adverse events(AEs) throughout VAD support per INTERMACS Definition
Time Frame: Six months and two years
Population: The number of subjects enrolled in the study and implanted with MVAD System.
Measure: Count of Participants; unit: Participants
Arm/Group | MVAD® Pump
Number analyzed (Participants) | 11
Participants
  Subjects with First Adverse Event by 6 months, cumulative. | 11
  Subjects with first Adverse Event by 2 years, cumulative. | 11

11. Secondary Outcome: Length of Initial Hospital Stay (Days)
Description: Length of Initial hospital stay (days) from procedure start to discharge
Time Frame: Post operation
Population: Subjects who underwent an MVAD implant attempt
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | MVAD® Pump
Number analyzed (Participants) | 11
Days | 40.2 (15.56)

12. Secondary Outcome: Re-Hospitalizations
Description: The length of Re-Hospitalization, excluding planned procedures, stay in days.
Time Frame: On or before 6 months follow-up and 24 month follow-up
Population: Subjects with an implant attempt
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | MVAD® Pump
Number analyzed (Participants) | 11
Days
  Length of Hospital Stay up to 6 month visit | 34.82 (110.22)
  Length of Hospital Stay Through 2 years | 69.91 (113.66)

13. Secondary Outcome: Transplantations
Description: Transplantations of subjects enrolled in study and implanted with MVAD System
Time Frame: Six months and two years
Population: The number of subjects enrolled in the study and implanted with MVAD System.
Measure: Count of Participants; unit: Participants
Arm/Group | MVAD® Pump
Number analyzed (Participants) | 11
Participants
  Subjects with transplant by 6 months, cumulative | 0
  Subjects with transplant by 2 years, cumulative | 3

14. Secondary Outcome: Explants
Description: Explants (i.e. death, transplant, recovery, device exchange) of MVAD in subjects enrolled in study and implanted with MVAD System
Time Frame: Six months and two years
Population: The number of subjects enrolled in the study and implanted with MVAD System.
Measure: Count of Participants; unit: Participants
Arm/Group | MVAD® Pump
Number analyzed (Participants) | 11
Participants
  Subjects with Explants by 6 months, cumulative | 1
  Subjects with Explants by 2 years, cumulative | 5

15. Secondary Outcome: New York Heart Association (NYHA) Functional Classification Score
Description: NYHA score measured at baseline, 6 month visit and 24 month visit. The NYHA scale is from I to IV. A subject with a score of IV indicates more severe heart failure than a subject with a score of I.
  Class I: No limitation of physical activity. Ordinary physical activity does not cause undue fatigue, palpitation or shortness of breath Class II: Slight limitation of physical activity. Comfortable at rest. Ordinary physical activity results in fatigue, palpitation, shortness of breath or chest pain Class III: Marked limitation of physical activity. Comfortable at rest. Less than ordinary activity causes fatigue, palpitation, shortness of breath or chest pain Class IV: Symptoms of heart failure at rest. Any physical activity causes further discomfort
Time Frame: Baseline and 6 month and 24 month visit
Population: Subjects implanted with MVAD
Measure: Count of Participants; unit: Participants
Groups:
- MVAD® Pump Baseline: Implant of HeartWare MVAD® System
  HeartWare MVAD® System: The HeartWare MVAD® System consists of a small, wearless, continuous flow pump and associated surgical tools and implant accessories, peripheral components which control and power the system, and a monitor which allows for programming and monitoring of the system
- MVAD Pump 6 Months: Subjects who underwent an implant attempt and had 6 month visit
- MVAD Pump at 24 Months: Subjects with MVAD pump implant attempt and 24 month visit
Arm/Group | MVAD® Pump Baseline | MVAD Pump 6 Months | MVAD Pump at 24 Months
Number analyzed (Participants) | 11 | 7 | 3
Participants
  Class I | 0 | 3 | 3
  Class II | 0 | 4 | 0
  Class III | 6 | 0 | 0
  Class IV | 5 | 0 | 0

16. Secondary Outcome: Length of Operative Time (Hours)
Description: Length of operative time (hours)
Time Frame: Implant
Population: Subjects who underwent an MVAD implant attempt
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | MVAD® Pump
Number analyzed (Participants) | 11
Hours | 2.78 (0.53)

ADVERSE EVENTS:
Time Frame: Through study completion: an average of 20.8 months but up to 2 years post implant.
Arm/Group | MVAD® Pump
All-Cause Mortality (participants affected / at risk) | 1/11
Serious Adverse Events (participants affected / at risk) | 7/11
Other Adverse Events (participants affected / at risk) | 10/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MVAD® Pump (N=11)
Arterial Non-CNS Thromboembolism (Vascular disorders) | 1 (1)
Cardiac Arrhythmia (Cardiac disorders) | 3 (4)
Device Malfunction/Failure (Product Issues) | 3 (7)
Hemolysis (Blood and lymphatic system disorders) | 4 (4)
Hepatic Dysfunction (Hepatobiliary disorders) | 1 (1)
Major Bleeding (Blood and lymphatic system disorders) | 7 (13)
Major Infection (Infections and infestations) | 3 (4)
Pericardial Fluid Collection (Cardiac disorders) | 2 (2)
Renal Dysfunction (Renal and urinary disorders) | 2 (2)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Other (General disorders) | 2 (11)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MVAD® Pump (N=11)
Cardiac Arrhythmias (Cardiac disorders) | 1 (1)
Device malfunction/failure (Product Issues) | 3 (3)
Major Infection (Infections and infestations) | 2 (3)
Other (General disorders) | 7 (27)

LIMITATIONS AND CAVEATS:
Due to the early suspension of enrollments, the target sample size of 57 was not reached. Fewer than 15 subjects were enrolled, thus no analysis was done.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2014-11-11): https://cdn.clinicaltrials.gov/large-docs/44/NCT01831544/Prot_000.pdf
  • Statistical Analysis Plan (2017-09-20): https://cdn.clinicaltrials.gov/large-docs/44/NCT01831544/SAP_001.pdf